CLINICAL TRIAL: NCT05238194
Title: Investigation Of The Psychological Effects of The Covid-19 Pandemic Process on The Health Staff Working in The Filation Team: A Mıxed Method Study
Brief Title: Psychological Effects of the Pandemic on the Health Personnel Working in the Filiation Team
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Associate Professor, Ordu University
Other Study IDs: Ordu12345
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Health Personnel
Keywords: Covid-19; Pandemic; Filiation; Health personnel; Psychological effect; Nursing; Trauma
MeSH Terms: conditions — COVID-19; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Psychological Effects of The Covid-19 Pandemic Process — Investigation of The Psychological Effects of The Covid-19 Pandemic Process on The Health Staff Workıng in The Filation Team

SUMMARY:
Purpose of Research: This study; It will be done in order to determine the psychological effects of the Covid-19 pandemic process on the health personnel working in the filiation team and to examine the possible effects in depth.

This research was planned as a mixed methods research. Research Questions

1. What are the psychological effects of the pandemic process on the healthcare personnel working in the filiation team?
2. Do the socio-demographic characteristics of the healthcare personnel working in the injection team affect their psychological status?
3. What are the opinions of the health personnel working in the filtering team about the psychological effects of the pandemic?

DETAILED DESCRIPTION:
Type of Research This research was planned as a mixed methods research. Mixed methods research is a type of research that allows us to obtain in-depth information from the data collected by quantitative and qualitative data collection techniques. It also defines it as a research approach in which quantitative and qualitative data are collected in order to understand research problems and two data sets are integrated with each other. In this approach, a better understanding of the problem is provided by combining statistical trends with stories and personal experiences (Yıldırım & Şimşek, 2011).

Research Pattern The design of this research was determined as an explanatory sequential mixed design, one of the mixed methods research designs. Creswell (2009) states that deciding on a mixed method design depends on four factors: timing (simultaneous-sequential), weight (qualitative-quantitative), when and how it is mixed (connected-integrative-embedded), and theorizing. In this study, the explanatory sequential mixed design, which is dependent on the timing factor, was adopted from the designs determined by Creswell and Plano Clark (2011). The purpose of adopting this design in the research is to explain the quantitative data to be collected in more depth with qualitative data. According to the exploratory sequential mixed design, in the research, first of all, the "Effect of Events Scale" will be applied to determine the psychological effects of the pandemic process on the healthcare personnel working in the filiation team, and then "Semi-Structured Interviews" will be conducted with questions to be prepared with the data obtained from the scale in order to investigate the reasons for the results from this scale. The exploratory sequential mixed pattern is shown as NIC nit. This pattern is expressed as a useful pattern when qualitative data are needed to explain quantitative results (Creswell & Guetterman, 2018).

ELIGIBILITY:
Inclusion Criteria:

* Worked in the filiation team,
* Open to communication and cooperation, and
* Healthcare personnel who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Healthcare personnel who worked during the filiation process but resigned due to various reasons such as retirement will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health personnel working in the filiation team
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale | 1.Day
  The scale developed by Weiss and Marmara (1997) was translated into Turkish by Çorapçıoğlu et al. (2006) Adapted by. The scale measures the subjective stress levels of individuals exposed to traumatic life events. The scale consists of 22 items, and each item is evaluated in a 5-point Likert type as (0) not at all, (1) a little, (2) moderate, (3) a lot, (4) a lot. A score between 0 and 88 is obtained from the scale, and a high score indicates that the person has a high level of post-traumatic stress disorder. The scale consists of three subscales: hyperarousal, avoidance, and re-experiencing. Reliving (questions 1, 2, 3, 6, 9, 14, 16, 20), Avoidance (questions 5, 7, 8, 11, 12, 13, 17, 22), and Overstimulation (4, 10, 15) , 18, 19, 21) are determined by these items.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Assoc. Dr., Principal Investigator — Ordu University
Locations (1):
- Hacer GOK UGUR, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No